CLINICAL TRIAL: NCT05691985
Title: Fibrinogen to Albumin Ratio (FAR) as a Risk Factor for Type 2 Diabetic Nephropathy(DN)
Brief Title: Fib to Alb Ratio in Type 2 Dkd
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdallah Gamal Abd El Hafeez Haridy, Resident, Assiut University
Other Study IDs: Fib to Alb ratio
Record Dates: First submitted 2023-01-11; First posted 2023-01-20 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: CKD; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aimed to investigate the association of fibrinogen to albumin ratio (FAR) with DKD type 2 and to prove its possible role as a novel biomarker to predict and prevent DKD progression.

DETAILED DESCRIPTION:
Diabetic kidney disease (DKD) is the most prevalent chronic kidney disease. Around 3540% of patients with type 2 diabetes mellitus (T2DM) will go on to develop DKD. DKD is characterized by albuminuria and reduced estimated glomerular filtration rate (eGFR), both of which are independent risk factors for end-stage kidney disease (ESKD), cardiovascular events, and death. DKD accounts for a significant increase in mortality among diabetic patients and is a grave threat to their clinical outcome.

Inflammation plays a major role in the development of DKD. Serum fibrinogen (FIB) is a biomarker of coagulation and inflammation. Elevated serum FIB is an independent risk factor of DKD progression to ESKD in patients with T2DM. Albumin (ALB) has anti-inflammatory functions and antioxidant properties. Hypoalbuminemia is associated with a poorer renal prognosis in patients with T2DM and DKD. Fibrinogen to albumin ratio (FAR) is a more significant prognostic marker than each single marker itself in cancer study.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 yrs.
* 50 Pts with type 2 DM that have DKD (presence of albuminuria in association with diabetic retinopathy) and 50 pts with type 2 DM but have no DKD.

Exclusion Criteria:

* Age below 18 yrs.
* Pts with ESKD, manifested cardiac valvular disease, acute infection, history of hepatitis, pts with DKA and Cancer.
* Pt who refused to contribute in this study

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients are selected on criteria of all genders, age above 18, type 2 DM and CKD. Patients are selected from clinics, community and pts admitted at hospital.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
The association of fibrinogen to albumin ratio (FAR) with DKD type 2. | baseline
  investigate the association of fibrinogen to albumin ratio (FAR) with DKD type 2.

CONTACTS AND LOCATIONS:
Overall Officials: Essam Abdelmonem Sadek, Prof, Study Director — Assiut University; Mohamed Hassan Mustafa, Dr, Study Director — Assiut University; Abdallah Gamal Abd El Hafeez, Resident, Principal Investigator — Assiut University

REFERENCES:
- [Background] Perez-Morales RE, Del Pino MD, Valdivielso JM, Ortiz A, Mora-Fernandez C, Navarro-Gonzalez JF. Inflammation in Diabetic Kidney Disease. Nephron. 2019;143(1):12-16. doi: 10.1159/000493278. Epub 2018 Oct 1. PMID 30273931
- [Background] GBD Chronic Kidney Disease Collaboration. Global, regional, and national burden of chronic kidney disease, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2020 Feb 29;395(10225):709-733. doi: 10.1016/S0140-6736(20)30045-3. Epub 2020 Feb 13. PMID 32061315
- [Background] Martinez-Castelao A, Navarro-Gonzalez JF, Gorriz JL, de Alvaro F. The Concept and the Epidemiology of Diabetic Nephropathy Have Changed in Recent Years. J Clin Med. 2015 May 28;4(6):1207-16. doi: 10.3390/jcm4061207. PMID 26239554
- [Background] Berhane AM, Weil EJ, Knowler WC, Nelson RG, Hanson RL. Albuminuria and estimated glomerular filtration rate as predictors of diabetic end-stage renal disease and death. Clin J Am Soc Nephrol. 2011 Oct;6(10):2444-51. doi: 10.2215/CJN.00580111. Epub 2011 Aug 18. PMID 21852671
- [Background] Luyendyk JP, Schoenecker JG, Flick MJ. The multifaceted role of fibrinogen in tissue injury and inflammation. Blood. 2019 Feb 7;133(6):511-520. doi: 10.1182/blood-2018-07-818211. Epub 2018 Dec 6. PMID 30523120
- [Background] Hsieh JY, Smith TD, Meli VS, Tran TN, Botvinick EL, Liu WF. Differential regulation of macrophage inflammatory activation by fibrin and fibrinogen. Acta Biomater. 2017 Jan 1;47:14-24. doi: 10.1016/j.actbio.2016.09.024. Epub 2016 Sep 20. PMID 27662809
- [Background] Zhang J, Wang Y, Zhang R, Li H, Han Q, Wu Y, Wang S, Guo R, Wang T, Li L, Liu F. Serum fibrinogen predicts diabetic ESRD in patients with type 2 diabetes mellitus. Diabetes Res Clin Pract. 2018 Jul;141:1-9. doi: 10.1016/j.diabres.2018.04.025. Epub 2018 Apr 21. PMID 29684616
- [Background] Zhang J, Zhang R, Wang Y, Li H, Han Q, Wu Y, Wang T, Liu F. The Level of Serum Albumin Is Associated with Renal Prognosis in Patients with Diabetic Nephropathy. J Diabetes Res. 2019 Feb 17;2019:7825804. doi: 10.1155/2019/7825804. eCollection 2019. PMID 30911552
- [Background] American Diabetes Association. 2. Classification and Diagnosis of Diabetes: Standards of Medical Care in Diabetes-2018. Diabetes Care. 2018 Jan;41(Suppl 1):S13-S27. doi: 10.2337/dc18-S002. PMID 29222373
- [Background] KDOQI. KDOQI Clinical Practice Guidelines and Clinical Practice Recommendations for Diabetes and Chronic Kidney Disease. Am J Kidney Dis. 2007 Feb;49(2 Suppl 2):S12-154. doi: 10.1053/j.ajkd.2006.12.005. No abstract available. PMID 17276798
- [Background] Sorensen I, Susnik N, Inhester T, Degen JL, Melk A, Haller H, Schmitt R. Fibrinogen, acting as a mitogen for tubulointerstitial fibroblasts, promotes renal fibrosis. Kidney Int. 2011 Nov;80(10):1035-44. doi: 10.1038/ki.2011.214. Epub 2011 Jul 6. PMID 21734641
- [Background] Myrup B, de Maat M, Rossing P, Gram J, Kluft C, Jespersen J. Elevated fibrinogen and the relation to acute phase response in diabetic nephropathy. Thromb Res. 1996 Feb 15;81(4):485-90. doi: 10.1016/0049-3848(96)00021-7. PMID 8907298
- [Background] Pan L, Ye Y, Wo M, Bao D, Zhu F, Cheng M, Ni X, Fei X. Clinical Significance of Hemostatic Parameters in the Prediction for Type 2 Diabetes Mellitus and Diabetic Nephropathy. Dis Markers. 2018 Feb 4;2018:5214376. doi: 10.1155/2018/5214376. eCollection 2018. PMID 29511389
- [Background] Tessari P, Kiwanuka E, Barazzoni R, Vettore M, Zanetti M. Diabetic nephropathy is associated with increased albumin and fibrinogen production in patients with type 2 diabetes. Diabetologia. 2006 Aug;49(8):1955-61. doi: 10.1007/s00125-006-0288-2. Epub 2006 May 16. PMID 16703327
- [Background] Erdogan G, Arslan U, Yenercag M, Durmus G, Tugrul S, Sahin I. Relationship Between the Fibrinogen-to-Albumin Ratio and SYNTAX Score in Patients with Non-St-Elevation Myocardial Infarction. Rev Invest Clin. 2021 Feb 3;73(3):182-189. doi: 10.24875/RIC.20000534. PMID 33535227